CLINICAL TRIAL: NCT04519385
Title: Toclizumam Versus Dexamethasone in Severe Covid-19 Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Alaa Rashad, Assistant professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SouthVU
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pneumonia, Viral
Keywords: COVID19; Tocilizumab; dexamethsone
MeSH Terms: conditions — Pneumonia, Viral; COVID-19 | interventions — tocilizumab; Dexamethasone

STUDY DESIGN:
Intervention Model Description: dexamethsone group Tocilizumab group
Who Masked: Participant, Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab
  Interventions: Drug: Tocilizumab
- Dexamethasone (Active Comparator): Dexamethasone therapy
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab therapy
  Other Names: TCZ
  Arms: Tocilizumab
Drug: Dexamethasone — dexamethsone pulse therapy
  Other Names: dexamethsone pulse therapy
  Arms: Dexamethasone

SUMMARY:
randomized controlled trial comparing survival benefit of Tocilizumab therapy with dexamethasone in patients with severe COVID 19

DETAILED DESCRIPTION:
The current study takes place in the ICU of ESNA hospital, the first COVID-19 quarantine hospital in Egypt, located in Upper Egypt, Luxor governorate during the period from March 2020 to June 2020.

The diagnosis of COVID-19 was made with a positive RT-PCR assay performed on a nasal swab. We have collected data on patients' demographics, comorbidities, symptoms, oxygen support, the ratio of partial pressure of arterial oxygen over the fraction of inspired oxygen (PaO2/FiO2 ratio), laboratory values (complete blood count, CRP, D-Dimer, ferritin, AST, ALT), diagnostic workup, therapies, complications, and outcomes.

Patients were given conventional treatment for COVID-19, including, hydroxychloroquine with a loading dose of 400 mg twice daily followed by 200 mg per day twice daily for additional five days and azithromycin 500 mg per day for five days unless contraindicated. An electrocardiogram was obtained for each patient to check the corrected QT interval at baseline.

In addition to conventional treatment, patients were randomly assigned to either dexamethasone group or tocilizumab (TCZ) group according to random tables.

Eligibility for study included patients with significant deterioration in respiratory clinical status with respiratory rate > 30 cycle/minute, Bilateral CT infiltration > 30%, PaO2/FiO2 ratio <150 or saturation <90 on >6L/min, Two positive laboratory tests of: (CRP>100 g/dL, lymphocytes<600 /mm3, D dimer>L, Ferritin >500).Interleukin 6 levels were not part of the criteria because it did not necessarily result in an actionable time frame.

Pediatric patients < 18 years old, patients with an active bacterial or fungal infection, and patients who were not requiring supplemental oxygen were excluded from the study.

No sample-size calculations were performed. The endpoint was time to failure, defined as death, within 14 days from ICU admission. Patients with a very early death reduced the risk that the treatment choice was motivated by the patient's disease course. Therefore, day 3 from hospital admission was set as a landmark time point: those who died, before the 3rd day of ICU admission, were excluded.

Treatment groups: Dexamethasone pulse therapy group:

All patients within this group received pulse Dexamethasone 4 mg/kg/day in an infusion form for the 3rd day, followed by a maintenance dose of 8 mg/day for 10 days with a subsequent withdrawal.

Tocilizumab group: Patients within this group received TCZ, 4 mg/kg/dose in 100 ccs normal saline over one hour. The same dose was repeated after 24h if there is no improvement in clinical assessment, corticosteroids (Solu-Medrol 40 mg for 5 days then 20 mg for 5 days) was added.

Data was collected at day one of treatment initialization, except for (PaO2/FiO2 ratio), which is also collected after 2 days from the end of the treatment and overall mortality within 14 days.

All patients provided informed consent for treatment with off label agents according to the local protocol approved by Hospital Authorities, for data collection and for participation in the study. The study was carried out in accordance with the principles of the Declaration of Helsinki and approved by the Regional Ethics Committee, Qena faculty of medicine, South-Vally University.

ELIGIBILITY:
Inclusion Criteria:

* respiratory rate > 30 cycle/minute, Bilateral CT infiltration > 30%, PaO2/FiO2 ratio <150 or saturation <90 on >6L/min, Two positive laboratory tests of: (CRP>100 g/dL, lymphocytes<600 /mm3, D dimer>L, Ferritin >500)

Exclusion Criteria:

* Pediatric patients < 18 years old, patients with active bacterial or fungal infection and patients who were not requiring supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Overall Survival at 14 days | 14 days
  survival 14 days from admission date

SECONDARY OUTCOMES:
Fio2/Pao2 | 2 days
  Change in Fio2/Pao2

CONTACTS AND LOCATIONS:
Overall Officials: Alaa R rashad, MD, Principal Investigator — South Valley University
Locations (1):
- Qena faculty medicine, Qina, Egypt